CLINICAL TRIAL: NCT06624150
Title: tDCS and Cognitive Training for Restrictive Eating Disorders
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: PSYCH-2022-31551
Record Dates: First submitted 2024-07-19; First posted 2024-10-02 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Anorexia Nervosa; Atypical Anorexia Nervosa
Keywords: anorexia nervosa; eating disorder; brain training; brain stimulation; fMRI
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Pilot mechanistic trial examining cognitive training and brain stimulation effects on cognitive performance. Participants are randomly assigned to active or sham (fake) brain stimulation conditions.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: triple blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active tDCS (Experimental): 10 Active tDCS sessions: 10 active sessions of transcranial direct current stimulation paired with cognitive training tasks. Device used is StarStim.
  Interventions: Device: Active tDCS sessions, StarStim device
- Sham (fake) tDCS (Sham Comparator): 10 Sham (fake) tDCS sessions: 10 fake sessions of transcranial direct current stimulation paired with cognitive training tasks. The device will be on the participants head, but the current will not be active.
  Interventions: Device: Sham (fake) tDCS sessions

INTERVENTIONS:
Device: Active tDCS sessions, StarStim device — 10 active sessions of transcranial direct current stimulation paired with cognitive training tasks. Device used is StarStim.
  Arms: Active tDCS
Device: Sham (fake) tDCS sessions — 10 fake sessions of transcranial direct current stimulation paired with cognitive training tasks. The device will be on the participants head, but the current will not be active.
  Arms: Sham (fake) tDCS

SUMMARY:
This study looks at adults with restrictive eating disorders who are currently receiving outpatient treatment for their eating disorder to examine whether a new brain stimulation technique called non-invasive transcranial direct current stimulation (tDCS) can enhance brain training. Participation involves interviews, assessments, 10 sessions of brain stimulation (active or sham), and computerized brain training over a 3-4 week period, with one post-intervention visit, and one 1-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Self-reported enrollment in outpatient-level treatment at local eating disorder treatment centers in the Twin Cities region, and meeting DSM-5 criteria for AN (mild severity, based on BMI greater than or equal to 17.0 kg/m2) or atypical AN diagnosis (based on MINI and EDE assessments).
* Participant must be capable of giving informed consent, based on UCSD Brief Assessment of Capacity to Consent (UBACC) risk assessment.
* Sufficient spoken English so as to be able to comprehend testing procedures. Normative ranges on a C-RENAL blood panel (panel and ranges specified here: https://labguide.fairview.org/showtest.asp?testid=3321)

Exclusion Criteria:

* Substance abuse in the participant
* Neurological condition or other developmental disorder
* Serious psychiatric disorder known to affect brain functioning and cognitive performance (e.g., schizophrenia, schizoaffective disorder)
* Medical instability, which will be evident based on required outpatient treatment status. In standard eating disorders treatment, individuals who are not medically stable are referred to higher levels of care (e.g., residential treatment, inpatient). Therefore, if a participant is enrolled in higher level care for their eating disorder diagnosis, this indicates medical instability and they will be excluded from enrollment in this study.
* tDCS contraindication (e.g., history of craniotomy, history of metallic cranial plates, screws, implanted devices).
* Acute suicidality (suicidalideation with a plan or intent), assessed via MINI suicidality module and Beck Depression Inventory suicide item
* Acute homicidality (homicidal ideation with a plan or intent), assessed via MINI
* Moderate, severe or extreme AN diagnostic severity, based on BMI as per DSM-5 criteria (e.g., BMI <17.0 kg/m2)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
the rate of dropout. | 14 days average
  Feasibility and tolerability measure 1. Evaluating for less than 20% dropout over the course of the tDCS for R-EDs study.
Number of participants retained in the tDCS | 14 days average
  Feasibility and tolerability measure 2 . # of participants retained in the tDCS and cognitive training space of the study (80% or more retention will be used as the assessment threshold).
probabilistic reversal learning task | 14 days average
  Change from pre intervention to post intervention scores in probabilistic reversal learning task performance
Dimensional set shifting task | 14 days average
  change from pre to post intervention scores in dimensional set shifting task.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Anderson, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States